CLINICAL TRIAL: NCT02518659
Title: Inulin- a Potential Preventive Dietary Supplement Against PPI Induced Hypomagnesemia
Brief Title: Prevalence and Intervention of Hypomagnesemia in Users of Proton-pump Inhibitors
Acronym: Privet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Joost Drenth, Professor, Radboud University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL nr.: 47262.091.13; NL37289.091.11 (Other: 2011/272)
Record Dates: First submitted 2015-06-26; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Hypomagnesemia, Intestinal, With Secondary Hypocalcemia; Drug Induced Hypomagnesemia
Keywords: hypomagnesemia; hypocalcemia; inulin; FOS; PPI; proton-pump inhibitors
MeSH Terms: conditions — Hypomagnesemia 1, Intestinal; Hypocalcemia | interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inulin (Other): Intervention by inulin, max 20gr per day
  Interventions: Dietary Supplement: Inulin
- No Inulin (No Intervention): Same Patients of arm inulin. Here the phase without inulin supplementation (own controls)

INTERVENTIONS:
Dietary Supplement: Inulin — This is the Intervention
  Other Names: Beneo Orafti Synergy1
  Arms: Inulin

SUMMARY:
Hypomagnesemia is a severe side effect of longterm use of all available proton-pump inhibitors (PPIH). It develops due to intestinal malabsorption of Mg2+.

This study investigates the application of dietary inulin fibers in users of proton-pump inhibitors with such a hypomagnesemia. To this end, repetitive short-term trials of 14 days of orally administered inulin, separated by a wash-out period of 14 days each were performed in cases of PPIH and controls. This study was not blinded or randomized.

DETAILED DESCRIPTION:
Hypomagnesemia due to PPI use (PPIH) has a low frequency, but is a difficult to control side effect in clinical practice. It develops over years and results in severe symptoms related to the hypomagnesemia. Due to the widespread use of PPIs, the real number of PPIH may be high. Currently, there is a lack of intervention strategies and no general treatment protocols for patients exist. It is generally anticipated that PPI-withdrawal and antacid replacement therapy is the only working method to recover patients from the hypomagnesemia. However, this frequently resulted in rebound of gastric acid related complaints.

The molecular mechanism of PPIH involves a reduction of Mg2+ absorption by the large intestine. Inulin fibers have been shown to have prebiotic properties. The intestinal microbiome ferments inulin and releases butyrate into the luminal compartment of the intestine. This results in acidification which enhances the uptake of Mg2+ and Ca2+ mediated by pH-sensitive ionchannels.Thus inulin may counteract PPI induced reduction of luminal protons and therefore reestablish normal Mg2+ absorption.

To this end cases with PPIH and controls underwent two 14 day trials of orally administered inulin under separated by wash-out periods of 14 days. During the experimental phase blood measures of electrolytes were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Chronic PPI use
* Hypomagnesemia

Exclusion Criteria:

* Uncontrolled diabetes
* Irregular use of the inulin fibers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cases and controls: Mean serum Mg2+ treatment effect of inulin (composite measure) | Cases and controls were followed for 56 days. Single measures of serum Mg2+ (in mmol/L) were performed at days 0, 14, 28,42 and 56.
  Measured values at respective timepoints are denoted as means +/- SEM in mmol/L. The treatment effect is calculated by the overall mean change of serum Mg2+ during the two inulin treated phases (Days 0 - 14 and days 28 - 42) and expressed as mean +/- SEM.

SECONDARY OUTCOMES:
Cases and controls: Mean serum Ca2+ treatment effect of inulin (composite measure) | Cases and controls were followed for 56 days. Single measures of serum Ca2+ (in mmol/L) were performed at days 0, 14, 28,42 and 56.
  Measured values at respective timepoints are denoted as means +/- SEM in mmol/L. The treatment effect is calculated by the overall mean change of serum Ca2+ during the two inulin treated phases (Days 0 - 14 and days 28 - 42) and expressed as mean +/- SEM.
Cases only: 24-hrs urine Mg2+ excretion without inulin at days 27/28 | Collected 24-hrs urine samples are taken from each case at days 27/28. Samples were stored and measured within one week after day 56, the finalizing day of the respective participant.
  Measured values for respective timepoint is denoted as a mean +/- SEM in mmol/24hrs.
Cases only: 24-hrs urine Mg2+ excretion with inulin at days 41/42 | Collected 24-hrs urine samples are taken from each case at days 41/42. Samples were stored and measured within one week after day 56, the finalizing day of the respective participant.
  Measured values for respective timepoint is denoted as a mean +/- SEM in mmol/24hrs.
Cases only: 24-hrs urine Ca2+ excretion without inulin at days 27/28 | Collected 24-hrs urine samples are taken from each case at days 27/28. Samples were stored and measured within one week after day 56, the finalizing day of the respective participant.
  Measured values for respective timepoint is denoted as a mean +/- SEM in mmol/24hrs.
Cases only: 24-hrs urine Ca2+ excretion with Inulin at days 41/42 | Collected 24-hrs urine samples are taken from each case at days 41/42. Samples were stored and measured within one week after day 56, the finalizing day of the respective participant.
  Measured values for respective timepoint is denoted as a mean +/- SEM in mmol/24hrs.
Cases and controls: General demographics of PPI users (Composite measure) | at day 0
  Demographical data, extracted from patient reports with relevant data such as age, sex, PPI-use and Duration and relevant comorbidities
Cases and Controls: Genetic screen of polymorphisms in the TRPM6 gene | DNA was extracted from blood, amplified and sequenced in average 2 months after bloodwithdrawal
  Small PCR and Sanger sequencing of exons 26+27 of the gene TRPM6 (Mg2+ channel)

CONTACTS AND LOCATIONS:
Overall Officials: René Bindels, Professor, Principal Investigator — Radboud University Medical Center

REFERENCES:
- [Background] Hess MW, Hoenderop JG, Bindels RJ, Drenth JP. Systematic review: hypomagnesaemia induced by proton pump inhibition. Aliment Pharmacol Ther. 2012 Sep;36(5):405-13. doi: 10.1111/j.1365-2036.2012.05201.x. Epub 2012 Jul 4. PMID 22762246
- [Background] Lameris AL, Hess MW, van Kruijsbergen I, Hoenderop JG, Bindels RJ. Omeprazole enhances the colonic expression of the Mg(2+) transporter TRPM6. Pflugers Arch. 2013 Nov;465(11):1613-20. doi: 10.1007/s00424-013-1306-0. Epub 2013 Jun 12. PMID 23756852
- [Background] Coudray C, Demigne C, Rayssiguier Y. Effects of dietary fibers on magnesium absorption in animals and humans. J Nutr. 2003 Jan;133(1):1-4. doi: 10.1093/jn/133.1.1. PMID 12514257